CLINICAL TRIAL: NCT03047096
Title: Intra-Articular, Single-shot Injection of Hyaluronic Acid and Corticosteroids in Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Dr. Shan-zheng Wang, Assitant secretory of Orthopaedics department, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZhongdaH2017
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis; Pain Syndrome; Intra-articular Injection
MeSH Terms: conditions — Osteoarthritis; Somatoform Disorders | interventions — Hyaluronic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA & CS group (Experimental): hyaluronic acid and corticosteroids
  Interventions: Drug: hyaluronic acid and corticosteroids
- HA group (Experimental): hyaluronic acid
  Interventions: Drug: hyaluronic acid

INTERVENTIONS:
Drug: hyaluronic acid — intra-Articular injection
  Other Names: HA
  Arms: HA group
Drug: hyaluronic acid and corticosteroids — intra-Articular injection
  Other Names: HA and CS
  Arms: HA & CS group

SUMMARY:
The aim of present study is to to investigate whether the combined injection of HA and CS was superior than HA alone in the treatment of knee OA.

DETAILED DESCRIPTION:
Intra-articular injection of hyaluronic acid (HA) or corticosteroids (CS) has been widely used with debate on its efficacy in osteoarthritis (OA). The aim of present study is to to investigate whether the combined injection of HA and CS is superior than HA alone in the treatment of knee OA.

ELIGIBILITY:
Inclusion Criteria:

According to radiographic findings, patients who are suffering from knee OA for over 3 months have to be stage II-IV according to the Kellgren-Lawrence (KL) grade by a senior radiologist. The diagnosis of symptomatic knee OA is based on American Rheumatism Association classification criteria for knee osteoarthritis.

Exclusion Criteria:

Exclusion criteria are the diagnosis of rheumatoid arthritis or other inflammatory OA, presence of trauma or pain-causing diseases, treatment with oral medications in recent 3 days, physiotherapy and intra-articular injection of HA or CS in the past 6 months. Participants who are allergic to any of the medications used in this study or diagnosed with current systemic infection are also excluded.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
VAS | 6 months
  Visual analog scale

SECONDARY OUTCOMES:
WOMAC | 6 months
  Western Ontario and McMaster University Osteoarthritis Index
Knee flexion motion | 6 months
  Knee flexion motion

CONTACTS AND LOCATIONS:
Overall Officials: Shan-zheng Wang, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No